CLINICAL TRIAL: NCT05762627
Title: Trajectories of Severe Eosinophilic Asthma During Childhood: Experience of the SAMP (Severe Asthma Molecular Phenotype) Cohort
Brief Title: Severe Eosinophilic Asthma Phenotypes During Childhood Have Various Origins
Acronym: SAMP 2
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220980
Record Dates: First submitted 2022-12-07; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Severe Asthma; Asthma in Children
Keywords: Childhood severe asthma; Eosinophilic asthma; Allergic asthma; Asthma trajectories; Type 2 inflammation
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of the clinical evolution at 10 years of children from the SAMP cohort (severe asthma, eosinophilic or not, allergic or not) in order to understand the different possible evolutions of these phenotypes at different ages.

DETAILED DESCRIPTION:
Multiple sensitizations but also blood eosinophilia are associated with the persistence of exacerbations during childhood. The pivotal role of eosinophilia in the pathophysiology of allergic asthma and more generally of severe asthma in the pediatric population has made it an important research topic for many years. The indirect demonstration of bronchial inflammation by analyzing blood eosinophilia is common practice, especially when monitoring the effectiveness of biotherapies. However, blood eosinophilia is not always clearly related to bronchial eosinophilia.

On the other hand, several teams have recently sought to highlight the recurrence of allergen sensitization profiles associated with severe asthma, in order to identify predictive factors of clinical evolution.

Finally, recent studies have shown that the nasal microbiota plays an important role in the onset, development and severity of asthma.

Our study will allow us to study the clinical evolution at 10 years of the children from the SAMP cohort (severe asthma, eosinophilic or not, allergic or not) in order to understand the different possible evolutions of these phenotypes at different ages. These phenotypic trajectories have an important therapeutic implication, leading to the prescription of personalized treatments, in particular biologics (monoclonal antibodies).

Primary objective To evaluate, in children with moderate to severe asthma, the control of asthma according to the therapeutic load, atopic pathologies during childhood and initial serum levels of blood eosinophils and biomarkers of eosinophil activation Secondary objective Evaluate the evolution of asthma phenotypes according to the associated atopic pathologies (allergic rhinitis, atopic dermatitis and food allergy), according to the number of atopic comorbidities and their severity.

Study of the microbiota in children followed for moderate to severe asthma.

Practical procedure The investigator record the new tests prescribed as part of the routine care of these patients (respiratory function tests, blood tests) and ask them to complete a questionnaire (no travel required specifically for the study). In the event of a blood test prescribed and carried out in the department, the investigator will take an additional 2 ml, and perform a nasal and skin swab.

ELIGIBILITY:
Inclusion Criteria:

* absence of opposition from the legal representative of the patient and if possible from the patient himself.
* patient with moderate to severe asthma at preschool or school age, previously included in SAMP Cohort

Exclusion Criteria:

* Patient included in another clinical study.
* Lack of coverage by social security.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from SAMP cohort
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
asthma control 1 | through study completion, 4 years
  Asthma control according to GINA (Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention, 2020. www.ginasthma.org.)
asthma control 2 | through study completion, 4 years
  Score of the Asthma Control Test (for children > 11 years old) and of the Asthma Control Test reserved for asthmatic children from 4 to 11 years old (ACT™, © 2002, by QualityMetric Incorporated Asthma France / French Control Test™ is a trademark of QualityMetric Incorporated. www.asthmacontroltest.com)

SECONDARY OUTCOMES:
asthma severity 1 | through study completion, 4 years
  Asthma severity according to GINA (Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention, 2022. www.ginasthma.org.)
asthma severity 2 | through study completion, 4 years
  Respiratory function tests (spirometry and plethysmography)
atopic comorbidities 1 | through study completion, 4 years
  Rhinitis control score: ARIA score (Allergic Rhinitis and its Impact on Asthma) endorsed by the WHO (Bousquet J, van Cauwenberge P, Khaltaev N, and the WHO panel members: Allergic Rhinitis and Its Impact on Asthma. ARIA. In collaboration with the World Health Organization. J Allergy Clin Immunol 2001; 108: S1-S315)
atopic comorbidities 2 | through study completion, 4 years
  Eczema control score: SCORAD score (Scoring atopic dermatitis) (Dermatology 1993; n°186 p23-p31. European Task Force of Atopic Dermatitis)
atopic comorbidities 3 | through study completion, 4 years
  Food allergy
nasal and skin microbiota | 1 day at inclusion of patient
  nasal and skin swabs for research of colonization with staphylococcus aureus

CONTACTS AND LOCATIONS:
Overall Officials: Mélisande Bourgoin-Heck, MD, MSc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Allergy Department, Trousseau Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided